CLINICAL TRIAL: NCT01289678
Title: Phase II Trial of Daily Pulse Interleukin-2 With Famotidine in Acute Myelogenous Leukemia
Brief Title: Trial of Daily Pulse Interleukin-2 With Famotidine in Acute Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to meet accrual goals
Sponsor: Leo W. Jenkins Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LJCC 06-05
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2017-03

CONDITIONS: Acute Myelogenous Leukemia
Keywords: acute myelogenous leukemia; interleukin-2
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Interleukin-2; Pulse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- interleukin-2 (Experimental): interleukin-2 therapy during lymphocyte recovery
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Famotine 20mg IV push daily just prior to the aldesleukin (IL-2) IL-2 18 million IU/m2 in 50 mL 5% D5 or NS IVPB over 15 - 30 minutes daily for 5 days
  Other Names: pulse

SUMMARY:
Assess the immunotherapy benefit of interleukin-2 in acute myelogenous leukemia treatment during lymphocyte recovery.

DETAILED DESCRIPTION:
Upon lymphocyte recovery after myeloablative induction standard chemotherapy pulse Interleukin-2 administered

ELIGIBILITY:
Inclusion Criteria:

* Confirmed hematopathology diagnosis of AML receiving marrow suppressive treatment
* Total WBC recovery of 500 mm3 prior to IL-2 treatment
* Platelet count of at least 20,000 mm3 prior to starting IL-2 treatment
* Active infection controlled prior to starting IL-2 treatment
* Stable systolic blood pressure > 90mm Hg prior to starting IL-2 treatment
* O2 saturation >90% prior to starting treatment
* Stable cardiopulmonary status prior to starting IL-2 treatment
* Serum creatinine < or equal to 2.0 mg/dl
* Total bilirubin and AST <3x upper limits normal

Exclusion Criteria:

* Acute Promyelocytic Leukemia
* Active thrombocytopenic bleeding
* Cardiac ejection fraction below 45%
* Pregnancy and/or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-07; Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Walker, MD, Principal Investigator — The Brody School of Medicine at East Carolina University
Locations (1):
- Leo W. Jenkins Cancer Center, Greenville, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interleukin-2
Started | 18
Completed | 12
Not Completed | 6
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | Interleukin-2
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 57 [32 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Event-free survival (EFS) = all patients; measured from the date of entry onto study until treatment failure, AML relapse, or death
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Interleukin-2
Number analyzed (Participants) | 12
Participants | 5

ADVERSE EVENTS:
Time Frame: 3 years post-consolidation therapy
Arm/Group | Interleukin-2
All-Cause Mortality (participants affected / at risk) | 7/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes